CLINICAL TRIAL: NCT04907019
Title: A Single Center, Open-label, Single Sequence Study to Evaluate the Potential Drug Interaction of CYP3A4 Inducer Rifampicin With SY-004 Capsules in Healthy Subjects
Brief Title: A Drug Interaction Study of SY-004 Capsules in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Suzhou Yabao Pharmaceutical R&D Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: SY004005
Record Dates: First submitted 2021-05-15; First posted 2021-05-28 (Actual); Last update posted 2022-05-18 (Actual); Status verified 2021-05

CONDITIONS: Type 2 Diabetes
Keywords: Drug interactions，rifampicin， Hypoglycemic drugs
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Group-drugs interaction (Experimental): 24 subjects were enrolled in this study. The effects of rifampicin single dose and steady-state on the pharmacokinetics of sy-004 will be analyzed.
  Interventions: Drug: rifampicin，SY-004

INTERVENTIONS:
Drug: rifampicin，SY-004 — On the morning of D1, the subjects will take orally 80 mg of SY-004 Capsules on an empty stomach.Fasting will be performed within 4 hours after taking the medicine. From D8 to D14, the subjects will take orally 600 mg rifampicin before breakfast every day. On the day of D15, the subjects will take orally 600 mg rifampicin and 80 mg SY-004 Capsules on an empty stomach.
  From D16 to D21, subjects will take orally 600 mg of rifampicin before breakfast every day.The patient can be discharged from the hospital after completing the safety examination on D22.

SUMMARY:
A single center, open-label, single sequence study was conducted to evaluate the potential drug interaction of CYP3A4 inducer rifampicin with SY-004 capsules in healthy subjects

ELIGIBILITY:
Inclusion Criteria:

* The subjects can communicate well with the researchers, understand and comply with the requirements of this study, and sign the informed consent voluntarily.
* Age on the day of signing the informed consent: healthy subjects aged 18 or above, both male and female.
* At the time of screening, male weight ≥ 50.0 kg, female weight ≥ 45.0 kg, 19.0 kg / m2 ≤ BMI ≤ 26.0 kg / m2.
* Fasting blood glucose ≥ 3.9 mmol / L and < 6.1 mmol / L.
* From one month before the informed consent to three months after the last medication, the subjects and their partners had no plans to have a child, take effective contraceptive measures voluntarily, and donate sperm or eggs.

Exclusion Criteria:

* Within 3 months before screening, a clinical trial was completed or withdrawn, or a clinical trial was in progress, or participated in other medical trial activities, and the researcher judged that it was not suitable to participate in this trial.
* With a history of serious systemic diseases or family history (including cardiovascular system, digestive system, urinary system, etc.), the researchers judged that the disease status could significantly change the absorption, distribution, metabolism and excretion of experimental drugs, or taking experimental drugs would increase the risk of subjects.
* Allergic constitution, or history of food allergy, or known allergy to study drug / similar drug, or to rifampicin or rifamycin antibiotics.
* Patients with previous orthostatic hypotension.
* Those who had a history of drug abuse, drug abuse or positive urine drug screening results in the past five years.
* Those who donated blood or lost more than 400ml in 4 weeks before screening, or received transfusion of blood or blood components in 4 weeks before screening, or planned to donate blood components within 3 months after the end of the study.
* Those who have a history of needle syncope or blood syncope, or who can't tolerate venipuncture for blood collection, or who have difficulty in blood collection.
* The patients with severe infection, trauma or major surgery within 4 weeks before the screening, or who plan to perform surgery during the study period (including but not limited to dental surgery).
* Use any prescription, over-the-counter, herbal or health products within 2 weeks before screening.
* Any drugs that inhibit or induce liver drug metabolizing enzymes were used within 30 days before screening.
* During the first three months of screening, the average alcohol intake was more than 14 units per week (1 unit = 360ml beer, 45ml spirits with 40% alcohol content or 150ml wine), or those who could not give up drinking during the test period, or those with positive alcohol breath.
* Smoking more than 5 cigarettes per day within 3 months before screening, or unwilling / unable to give up smoking during the trial.
* Those who have special requirements for diet and can not comply with the unified diet arrangement.
* It is not guaranteed that chocolate, any food or drink containing caffeine or possibly affecting the test results (such as pitaya, grapefruit, grapefruit, orange juice, mango, etc.) will be fasted 48 hours before administration and during the test.
* Pregnant or lactating women, or pregnancy test results were positive.
* The screening results of HBsAg, HCV, TP and HIV were positive.
* When screening, there was ALT > 1.5 times the upper limit of normal value（ × ULN), or ast > 1.5 × ULN, or TBIL > 1.5 × ULN。
* When screening, the 12 lead ECG showed the following results: QT interval (qtcb) > 450ms (male) or > 470ms (female).
* The results of physical examination, vital signs, abdominal B-ultrasound (liver, gallbladder, pancreas, spleen and kidney), chest CT, ECG, laboratory examination items and test related auxiliary examination in screening period were not suitable for the participants.
* According to the judgment of the researcher, the subjects with other factors not suitable to participate in the experiment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2021-07-06 (Actual); Primary Completion 2021-08-17 (Actual); Study Completion 2021-08-17 (Actual)

PRIMARY OUTCOMES:
Cmax | 22 days
  Peak Plasma Concentration (Cmax) of SY-004 when SY-004 capsules were treated with rifampicin alone or in combination with rifampicin at steady-state level
AUC0-t | 22 days
  Area under the plasma concentration versus time curve (AUC0-t)) of SY-004 when SY-004 capsules were treated with rifampicin alone or in combination with rifampicin at steady-state level
AUC0-∞ | 22 days
  Area under the plasma concentration versus time curve (AUC0-∞)) of SY-004 when SY-004 capsules were treated with rifampicin alone or in combination with rifampicin at steady-state level

SECONDARY OUTCOMES:
Tmax | 22 days
  Peak Time （Tmax）of SY-004 when SY-004 capsules were treated with rifampicin alone or in combination with rifampicin at steady-state level
T1/2z | 22 days
  Half time （T1/2z）of SY-004 when SY-004 capsules were treated with rifampicin alone or in combination with rifampicin at steady-state level
CLz/F | 22 days
  Clearance (Clz/F)of SY-004 when SY-004 capsules were treated with rifampicin alone or in combination with rifampicin at steady-state level

CONTACTS AND LOCATIONS:
Locations (1):
- XIE Haitang, Wuhu, Anhui, China